CLINICAL TRIAL: NCT04385290
Title: MidOStaurin + Gemtuzumab OzogAmIcin Combination in First-line Standard Therapy for Acute Myeloid Leukemia (MOSAIC)
Brief Title: Combination of Midostaurin and Gemtuzumab Ozogamicin in First-line Standard Therapy for Acute Myeloid Leukemia (MOSAIC)
Acronym: MOSAIC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUD-MOSAIC-075
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; FLT3 mutation; CBF; midostaurin; gemtuzumab ozogamicin
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — midostaurin; Gemtuzumab

STUDY DESIGN:
Intervention Model Description: The phase I dose escalation trial (MODULE) will be conducted according to the 3+3 design.
  The phase II trial in CBF AML (MAGNOLIA) will be conducted in a open label and randomized manner.
  The phase II trial in FLT3 mutated AML (MAGMA) will be conducted in a open label and randomized manner.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subtrials are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MODULE trial: dose escalation (Experimental): Phase I (Trial part MODULE): The treatment plan combines increasing doses levels of midostaurin (25/50 mg BID) and gemtuzumab ozogamicin (3 mg/m^2 i.v. max 4.5 mg on day(s) 1, (4, 7)) with 7+3 standard chemotherapy scheme using cytarabine (200 mg/m^2 cont. inf. i.v. on days 1 to 7) and daunorubicin (60 mg/m^2 i.v. on days 1 to 3).
  Interventions: Drug: MODULE: conventional chemotherapy (Cytarabine+Daunorubicin) in combination with midostaurin+GO
- MAGNOLIA-trial: conventional chemotherapy+GO and midostaurin (Experimental): Phase II (Trial part MAGNOLIA): midostaurin (recommended phase II dose, RP2D) is combined with treatment standard (7+3 standard chemotherapy scheme using cytarabine 200 mg/m^2 cont. inf. i.v. and daunorubicin 60 mg/m^2 i.v.) plus GO (recommended phase II dose, RP2D) in CBF AML
  Interventions: Drug: MAGNOLIA-trial: Midostaurin associated with conventional chemotherapy (AraC+DNR)+GO
- MAGNOLIA-trial: conventional chemotherapy+GO (Active Comparator): Phase II (Trial part MAGNOLIA): treatment standard of CBF AML (7+3 standard chemotherapy scheme using cytarabine 200 mg/m^2 cont. inf. i.v. and daunorubicin 60 mg/m^2 i.v. plus GO (3 mg/m^2 i.v. max 4.5 mg) on days 1, 4, 7). No additional Midostaurin is given.
  Interventions: Drug: MAGNOLIA-trial: conventional chemotherapy (AraC+DNR)+GO
- MAGMA-trial: conventional chemotherapy+midostaurin and GO (Experimental): Phase II (Trial part MAGMA): GO (recommended phase II dose, RP2D) is combined with treatment standard (7+3 standard chemotherapy scheme using cytarabine 200 mg/m^2 cont. inf. i.v. and daunorubicin 60 mg/m^2 i.v.) plus Midostaurin (recommended phase II dose, RP2D) in FLT3 mutated AML
  Interventions: Drug: MAGMA-trial:GO associated with conventional chemotherapy (AraC+DNR)+Midostaurin
- MAGMA-trial: conventional chemotherapy+midostaurin (Active Comparator): Phase II Trial (MAGMA): treatment standard of FLT3 mutated AML (7+3 standard chemotherapy scheme using cytarabine 200 mg/m^2 cont. inf. i.v. and daunorubicin 60 mg/m^2 i.v plus midostaurin). No additional GO is given.
  Interventions: Drug: MAGMA-trial: conventional chemotherapy (AraC+DNR)+Midostaurin

INTERVENTIONS:
Drug: MODULE: conventional chemotherapy (Cytarabine+Daunorubicin) in combination with midostaurin+GO — Midostaurin (IMP) induction: 25 mg or 50 mg peroral BID, days 8 to 21 depending on assigned dose level
  GO (IMP) induction: 3 mg/m^2 i.v. max 4.5 mg, on day1, or on days 1, 4, or days 1, 4, 7 depending on assigned dose level
  Daunorubicin (DNR, non-IMP) induction: 60 mg/m^2/day i.v., days 1 to 3
  Cytarabine (AraC, non-IMP) induction: 200 mg/m^2/day cont. infusion, days 1 to 7
  Other Names: Rydapt; Mylotarg
  Arms: MODULE trial: dose escalation
Drug: MAGNOLIA-trial: Midostaurin associated with conventional chemotherapy (AraC+DNR)+GO — Midostaurin (IMP):
  RP2D peroral, days 8 to 21, induction cycle 1; 50 mg peroral BID, days 8 to 21 induction cycle 2; 50 mg peroral BID, days 8 to 21, 3 consolidation cycles; 50 mg peroral BID, days 1 to 28, 12 maintenance cycles;
  GO (IMP): 3 mg/m^2 i.v. max 4.5 mg, RP2D, 1 induction cycle only
  Daunorubicin (DNR, non-IMP):
  60 mg/m^2 i.v., days 1 to 3 of induction cycle 1 and 2 in good and moderate responders; 50 mg/m^2/day i.v., days 1 to 3 of induction cycle 2 in non-responders
  Cytarabine (AraC, non-IMP):
  200 mg/m^2/day cont. infusion, days 1 to 7 of induction cycles 1 and 2 in good and moderate responders; 3000/1500 mg/m^2/day i.v. BID, days 1 to 3 of induction cycle 2 in non-responders; 3000/1500 mg/m^2 i.v. BID, days 1, 3, 5 of consolidation, 3 cycles
  Other Names: Rydapt; Mylotarg
  Arms: MAGNOLIA-trial: conventional chemotherapy+GO and midostaurin
Drug: MAGNOLIA-trial: conventional chemotherapy (AraC+DNR)+GO — GO (IMP): 3 mg/m^2 i.v. max 4.5 mg on days 1, 4, 7; 1 induction cycle only
  Daunorubicin (DNR, non-IMP):
  60 mg/m^2/day i.v., days 1 to 3 of induction cycle 1 and 2 in good and moderate responders; 50 mg/m^2/day i.v., days 1 to 3 of induction cycle 2 in non-responders
  Cytarabine (AraC, non-IMP):
  200 mg/m^2/day cont. infusion, days 1 to 7 of induction cycles 1 and 2 in good and moderate responders; 3000/1500 mg/m^2/day i.v. BID, days 1 to 3 of induction cycle 2 in non-responders; 3000/1500 mg/m^2 i.v. BID, days 1, 3, 5 of consolidation, 3 cycles
  Other Names: Mylotarg
  Arms: MAGNOLIA-trial: conventional chemotherapy+GO
Drug: MAGMA-trial:GO associated with conventional chemotherapy (AraC+DNR)+Midostaurin — Midostaurin (IMP):
  RP2D peroral, days 8 to 21, induction cycle 1; 50 mg peroral BID, days 8 to 21, induction cycle 2; 50 mg peroral BID, days 8 to 21, 3 consolidation cycles; 50 mg peroral BID, days 1 to 28, 12 maintenance cycles;
  GO (IMP): 3 mg/m^2 i.v. max 4.5 mg, RP2D, 1 induction cycle only
  Daunorubicin (DNR, non-IMP):
  60 mg/m^2/day i.v., days 1 to 3 of induction cycles 1-2 in good and moderate responders; 50 mg/m^2/day i.v., days 1 to 3 of induction cycle 2 in non-responders
  Cytarabine (AraC, non-IMP):
  200 mg/m^2/day cont. infusion, days 1 to 7 of induction cycles 1 and 2 in good and moderate responders; 3000/1500 mg/m^2/day i.v. BID, days 1 to 3 of induction cycle 2 in non-responders; 3000/1500 mg/m^2 i.v. BID, days 1, 3, 5 of consolidation, 3 cycles
  Other Names: Mylotarg; Rydapt
  Arms: MAGMA-trial: conventional chemotherapy+midostaurin and GO
Drug: MAGMA-trial: conventional chemotherapy (AraC+DNR)+Midostaurin — Midostaurin (IMP):
  RP2D peroral, days 8 to 21, induction cycle 1; 50 mg peroral BID, days 8 to 21 induction cycle 2; 50 mg peroral BID, days 8 to 21, 3 consolidation cycles; 50 mg peroral BID, days 1 to 28, 12 maintenance cycles
  Daunorubicin (DNR, non-IMP):
  60 mg/m^2/day i.v., days 1 to 3 of induction cycle 1 and 2 in good and moderate responders; 50 mg/m^2/day i.v., days 1 to 3 of induction cycle 2 in non-responders
  Cytarabine (AraC, non-IMP):
  200 mg/m^2/day cont. infusion, days 1 to 7 of induction cycles 1 and 2 in good and moderate responders; 3000/1500 mg/m^2/day i.v. BID, days 1 to 3 of induction cycle 2 in non-responders; 3000/1500 mg/m^2 i.v. BID, days 1, 3, 5 of consolidation, 3 cycles
  Other Names: Rydapt
  Arms: MAGMA-trial: conventional chemotherapy+midostaurin

SUMMARY:
This phase I/II clinical trial evaluates the safety and efficacy of the combined administration of midostaurin and gemtuzumab ozogamicin in the frame of first-line standard chemotherapy in newly diagnosed acute myeloid leukemia (AML) patients displaying a cytogenetic aberration or fusion transcript in the core-binding factor (CBF) genes or FMS-like tyrosine Kinase 3 (FLT3) mutation.

DETAILED DESCRIPTION:
Acute myeloid leukemia is a malignancy that is still fatal for the majority of patients. Besides age, the genetic configuration of AML blasts is one of the strongest prognostic factors. Patients with mutations in the core-binding factor (CBF) genes have the best prognosis, however a considerable proportion of 35-60% will eventually relapse. Mutation and overexpression of receptor tyrosinkinases (RTK) have been proposed as main reasons for relapse development or chemoresistance in CBF AMLs. RTKs like stem cell factor receptor (c-KIT) and FLT3 are of high clinical relevance as they mediate proliferation and differentiation of hematopoietic stem cells. There is evidence that c-Kit mutations and high levels of c-KIT in CBF-AML have adverse effects on survival endpoints indicating c-KIT as potential therapeutic target in this special AML population. Midostaurin can be considered a potent c-KIT inhibitor besides having multi-kinase inhibitory activity for several other kinases of documented or potential pathogenetic relevance for AML, most importantly mutated FLT3. The kinase inhibition ultimately leads to inhibition of proliferation, cell cycle arrest, and apoptosis. Previous studies with other c-KIT inhibitors such as dasatinib showed promising results with respect to survival end points in newly diagnosed CBF AML patients. Midostaurin is considered a more potent c-KIT inhibitor than dasatinib and may be able to potentiate the inhibitory effect on leukemic cell growth.

Another important therapeutical target in CBF AML is the sialic acid-binding immunoglobulin-like lectin (CD33) which is expressed on the majority of AML blasts. Gemtuzumab Ozogamicin (GO) is a therapeutic CD33 antibody linked to a strong cytostatic drug (calicheamicin) which causes apoptosis of cancer cells upon internalization. For the combination of GO and standard intensive chemotherapy, metaanalyses of randomized trials have shown that i) a low-dose fractionated administration results in the best tolerability, and ii) among AML subgroups, patients with CBF AML have the greatest benefit from GO in addition to standard therapy. Subgroup analyses within the ALFA-0701 (A Randomized Study of Gemtuzumab Ozogamicin With Daunorubicine and Cytarabine in Untreated Acute Myeloid Leukemia Aged of 50-70 Years Old) trial population showing beneficial effects of GO on overall survival, relapse-free survival and event-free survival in patients positive for FLT3 mutation as compared to those negative for FLT3 mutation. Subgroup analyses of the GO registration trial ALFA-0701 showed a significant clinical benefit of the patients displaying a mutation in the FLT3 gene compared to those without this mutation. In Addition, CBF AML patients with FLT3 mutations expressed particularly high levels of CD33 antigen and that CD33 antigen levels were positively correlated to the improved survival after GO treatment. Furthermore, recently published data of two paediatric populations with internal tandem mutation in the FLT3 gene showed reduced relapse rates in GO recipients compared to the control group only receiving standard chemotherapy. These results suggest that GO is a particularly beneficiary agent in FLT3 mutated patients who would currently receive midostaurin in addition to intensive chemotherapy as a standard of care. Hence, from a clinical point of view there is an unambiguous rationale supporting the combination of midostaurin and GO for treatment of AML in the two cytogenetic subgroups: CBF AML and FLT3 mutated AML.

GO has become the new treatment standard for patients with CBF AML. The hypothesized positive effect of midostaurin is likely but randomized proof is laking.

Midostaurin has become the new treatment standard for AML patients with mutations in the FLT3 gene. The positive effect of GO is shown in a post-hoc subgroup analysis of the ALFA-0701 trial, but prospective randomized proof is lacking.

Therefore, the proposed trial intends i) to explore and establish the safe combination of GO plus midostaurin (MODULE) and ii) to evaluate the effect of midostaurin versus no midostaurin added to standard AML chemotherapy plus GO in CBF AML (MAGNOLIA) and iii) to evaluate the effect of GO versus no GO added to standard AML chemotherapy plus midostaurin in FLT3 mutated AML (MAGMA).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Newly diagnosed AML according to the criteria of the World Health Organisation plus the following molecular or cytogenetic specifications:

  * Phase I Trial - MODULE:

    * t(8;21)/RUNX1-RUNX1T1 or
    * inv(16) or t(16;16)/CBFB-MYH11 or
    * FLT3-ITD or
    * FLT3-tyrosine kinase domain (FLT3-TKD)
  * Phase II Trial - MAGNOLIA

    * t(8;21)/RUNX1-RUNX1T1 or
    * inv(16) or t(16;16)/CBFB-MYH11
  * Phase II Trial - MAGMA

    * FLT3-ITD or
    * FLT3-TKD
    * Absence of mutations in CBF genes (i.e. t(8;21)/RUNX1-RUNX1T1 or inv(16) or t(16;16)/CBFB-MYH11)
* Male and female patients aged

  * 18 - ≤ 75 years in Phase I Trial - MODULE
  * 18 - ≤ 70 years in Phase II Trials - MAGMA and MAGNOLIA
* Eastern Cooperative Oncology Group (ECOG) Score of 0-2
* Life expectancy > 14 days
* Adequate hepatic and renal function

  * alanine aminotransferase / aspartate transaminase ≤ 2.5 x ULN
  * Bilirubin < 2 x upper limits of normal
  * Creatinine < 1.5 x upper limits of normal or Creatinine clearance > 40 ml/min
* White blood cell count < 30 × 10^9/L. Note: Hydroxyurea and/or a dose of 100-200 mg/m^2 cytarabine per day for up to 3 days (for emergency use for clinical stabilization) is permitted to meet this criterion.

Exclusion Criteria (all study parts):

* Previous antineoplastic treatment for AML other than hydroxyurea and/or cytarabine for emergency use (100-200 mg/m^2 per day on maximal 3 days)
* Previous treatment with anthracyclines
* central nervous system involvement
* Isolated extramedullary AML
* Uncontrolled infection
* AML after antecedent myelodysplasia (MDS) with prior cytotoxic treatment (e.g., azacytidine or decitabine)
* Any investigational agent within 30 days or 5 half-lives, whichever is greater, prior to day 1. An investigational agent is defined as an agent with no approved medical use in adults or in pediatric patients
* Prior treatment with a FLT3 inhibitor (e.g., midostaurin, quizartinib, sorafenib)
* Strong CYP3A4/5 enzyme inducing drugs unless they can be discontinued or replaced prior to enrollment
* Any other known disease or concurrent severe and/or uncontrolled medical condition (e.g., cardiovascular disease including congestive heart failure or active uncontrolled infection) that could compromise participation in the study
* Impairment of gastrointestinal (GI) function or GI disease that might alter significantly the absorption of midostaurin
* Confirmed diagnosis of HIV infection,
* Active viral hepatitis unless serology demonstrates clearance of infection. Occult or prior hepatitis B virus (HBV) infection, defined as negative hepatitis B surface antigen and positive total hepatitis core antibodies, may be included if HBV DNA is undetectable, provided that patients are willing to undergo monthly DNA testing. Patients who have protective titers of hepatitis B surface antibody after vaccination or prior cured hepatitis B are eligible. Patients for hepatitis C virus (HCV) antibody are eligible provided PCR is negative for HCV RNA.
* Cardiovascular abnormalities, including any of the following:

  * History of myocardial infarction, angina pectoris, Coronary Artery Bypass Grafting within 6 months prior to starting study treatment
  * Clinically uncontrolled cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular block (e.g., bifascicular block, Mobitz type II and third degree atrioventricular block)
  * Uncontrolled congestive heart failure
  * Left ventricular ejection fraction of < 50%
  * Poorly controlled arterial hypertension
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they fulfill at least one of the following criteria:

  * Post-menopausal (12 months of natural amenorrhea or 6 months of amenorrhea with serum follicule stimulating hormone > 40 U/ml)
  * Postoperative (i.e. 6 weeks) after bilateral ovariectomy with or without hysterectomy
  * Women of childbearing potential must have a negative serum pregnancy test performed within 7 days before the first dose of study drug
  * Continuous and correct application of a contraception method with a Pearl Index of < 1% (e.g. implants, depots, oral contraceptives, intrauterine device) from initial study drug administration until at least 7 months after the last dose of gemtuzumab ozogamicin and at least 4 months after the last dose of midostaurin, whichever period is longer. A hormonal contraception method must always be combined with a barrier method (e.g. condom)
  * Sexual abstinence
  * Vasectomy of the sexual partner
* Sexually active males unless they use a condom during intercourse while taking the drug during treatment, and for at least 4 months after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via semen
* Unwillingness or inability to comply with the protocol
* Known hypersensitivity to midostaurin, GO, cytarabine or daunorubicin or to any of the excipients of midostaurin, GO, cytarabine or daunorubicin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of midostaurin and GO combination | treatment day 8 until day 42 at the latest
  as measured by the number of dose limiting toxicities related to midostaurin or GO exposure.
Event Free Survival (EFS) | up to 3 years from enrolment
  Time interval from date of randomization until either primary treatment failure or relapse or death, whichever occurs first.

SECONDARY OUTCOMES:
CR/CRi rate | after induction treatment, approx. 2 months
  CR/CRi rate is defined as the proportion of patients, who achieved a morphologic complete remission or a complete remission with incomplete hematologic recovery (CR or CRi) during study participation.
Duration of remission | up to 3 years from enrolment
  Duration of remission is defined as time interval from date of CR/CRi until morphologic relapse.
Cumulative incidence of relapse | up to 3 years from enrolment
  Cumulative incidence of relapse is defined as the time interval from date of first CR/CRi until relapse.
Relapse-free survival | up to 3 years from enrolment
  Relapse-free survival is defined as the time interval from date of first CR/CRi until either morphologic relapse or death in remission.
Overall survival | up to 3 years from enrolment
  Overall survival is defined as time interval from date of randomization until death from any cause.
Early mortality rate | 30 and 60 days after commencement of therapy
  Early mortality is defined as death from any reason within 30 days and 60 days from start of induction.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Röllig, Prof. Dr., Principal Investigator — Technische Universität Dresden, Medical Faculty Carl Gustav Carus
Locations (21):
- Germany (21):
  - LMU Klinikum, Campus Großhadern, München, Bavaria
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Aachen, Aachen
  - Universitätsklinikum Augsburg, Augsburg
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum Dresden, Dresden
  - Johann Wolfgang Goethe-Universität, Frankfurt am Main
  - Universitätsklinikum Halle, Halle
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Gemeinschaftsklinikum Mittelrhein gGmbH, Koblenz
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Mannheim gGmbH, Mannheim
  - Philipps-Universität Marburg Fachbereich Medizin, Marburg
  - Rotkreuzklinikum München gGmbH, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg-Nord, Nuremberg
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Rems-Murr-Klinikum Winnenden, Winnenden

REFERENCES:
- See also: homepage of study group — https://www.aml-germany.com